CLINICAL TRIAL: NCT05503745
Title: CBT-E vs CBT-F+Metacognitive Interpersonal Therapy for Non-underweight Adults With Eating Disorders: Study Protocol for a Pilot Randomised Controlled Trial
Brief Title: MICBT for Non-underweight Adults With Eating Disorders
Acronym: MICBT-ED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Trattamento Integrato: Disturbi Alimentari e Obesita (Other)
Responsible Party: Principal Investigator, GLORIA FIORAVANTI, Psychotherapist, Centro Trattamento Integrato: Disturbi Alimentari e Obesita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000781
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Eating Disorders; Maladaptive Personality Trait; Emotion Regulation; Personality; Personality Disorders; Social Interaction; Perfectionism; Self Esteem; Cognitive Dysfunction; Dysfunctional Behavior, Psychology
MeSH Terms: conditions — Feeding and Eating Disorders; Emotional Regulation; Personality Disorders; Cognitive Dysfunction; Problem Behavior

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized controlled trial design will be used in order to compare CBT-E (n = 10) condition to combined MIT/CBT-F (n = 10). Patients in both conditions will receive 20 weekly sessions of either CBT-E or CBT-F+MIT. Repeated follow-up will be collected up to 24 months. The study is run in an private outpatient clinic specialized in eating disorder treatment. We will evaluate acceptability in terms of session attendance and number of completers and preliminary outcomes.
Who Masked: Outcomes Assessor
Masking Description: Each participant will be randomized in one of the two experimental conditions by allocation concealment. In particular, randomized-permuted blocks will be used. The research team will be also blind to the randomized allocation. Group allocation will remain concealed until the end of the assessment stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-E (Active Comparator): Participants in the CBT-E condition will receive a total of 20 CBT-E sessions over 20 weeks. CBT-E treatment will consist of four stages. In particular, CBT aims to inform patients about the importance of self-control, the dangers of some restrictive behaviors such as self-induced vomiting. Moreover, CBT provides strategies to patients in order to monitor their usually dysfunctional behaviors and so increasing their awareness (i.e. food diary method) while reducing the availability of food and encourages activities that are incompatible with overeating. Patients will be trained in problem solving in order to change these feelings, as well as in increasing their self-awareness in order to recognize irrational thoughts about their body weight and shape. Additionally, they will be gradually exposed to foods that they had been avoiding.
  Interventions: Other: CBT-E
- CBT-F+MIT (Experimental): Participants in the CBT-F+MIT condition will receive a total of 20 sessions over 20 weeks. Specifically, 2 sessions will be based on CBT-F as usual only. During these sessions participants will receive psychoeducational training on eating behaviors and an introduction to the protocol tools, namely the monitoring form, weight chart, transdiagnostic formulation and Eating Problem Check List (EPCL).
  These elements will be used at the beginning of the remaining 18 sessions, in order to monitor the regulations of eating behaviors as well eliciting narrative episodes. These materials will form the basis for the MIT-part of the session, in which therapists will seek to form with the patient a shared understanding of the psychological reasons underlying their ED symptoms and their maladaptive interpersonal functioning. MIT sessions will be integrated within the CBT-F protocol which will provide psycho-educational, nutritional re-education and management for ED.
  Interventions: Other: CBT-F+MIT

INTERVENTIONS:
Other: CBT-F+MIT — The aim is to develop healthier strategies for managing negative thoughts and feelings antecedent to ED and for engaging patients in social interactions that meet their relational basic wishes. They will thus understand that perfectionism and the need for control they experience through ED are coping strategies developed within interpersonal patterns of interaction with significant others, where low self-esteem and emotive dysregulation play a central role. MIT aims to improve individuals' capacity to make sense of their own affect and cognitions and become aware of being driven by maladaptive, rigid and biased schemas about self and others, to form a richer understanding of the mind of the others and use this knowledge to react in more adaptive ways to social difficulties or evolutionary selected wishes. MIT also enables individuals to reflect on how these schemas may act as triggers for ED behavior and to develop more effective coping strategies in face of interpersonal stressors.
  Arms: CBT-F+MIT
Other: CBT-E — In the first Stage, the treatment will be focused on achieving a shared understanding of the patient's eating disorder and the related maintenance factors. In this phase the patient will be helped to regulate and stabilize his eating habits and so to address his weight concerns. In the second stage, progress made is reviewed in detail. In the third stage, the sessions will be focused on the central processes that are maintaining the psychopathology of the patient's eating disorder. In particular, this involves in addressing concerns about weight and body shape, cognitive and caloric dietary restriction, events and emotions that affect nutrition. In phase three and four clinical perfection, low global self-esteem, intolerance of emotions and interpersonal difficulties are also addressed. Towards the end of the third stage and during the fourth stage, procedures will be also implemented to minimize the risk of short- and long-term relapse.
  Arms: CBT-E

SUMMARY:
Eating disorders (ED) are severe but treatable conditions, but there are large margin for improvements in terms of efficacy and adherence. There is room to explore new treatment options who are either more capable to retain patients in therapy, more effective. Alternative their efficacy may match the ones of current available treatments but offer new options to ones that did not respond to available therapies. Here the investigators explored if a combination of CBT-focused plus Metacognitive Interpersonal Therapy (MIT) is an empirically supported therapy for personality disorders and could be a new viable treatment option for non-underweight ED. MIT targets some aspects of ED such as poor awareness of mental states and maladaptive interpersonal schemas that are not included in the transdiagnostic model underlying the most investigated empirically supported treatment for ED that is CBT-E. It is reasonable therefore that targeting these aspects of psychopathology can be a path to treatment adherence and effectiveness

DETAILED DESCRIPTION:
The study is a pilot randomized controlled trial that aims to evaluate the feasibility and effectiveness of weekly MIT in addiction to CBT-F in a group of adults diagnosed with ED. Specifically, the investigators will investigate in a sample of non-underweight adults presenting with ED whether once compared to CBT-E, a treatment combining MIT and CBT-F is a) feasible, b) well-tolerated and c) potentially effective on eating disorders symptoms and other outcomes.

The investigators expect that the experimental group CBT-F+MIT would be able to have high treatment adherence and retention on the ground of previous studies of MIT for personality disorders. They will also expect good outcomes in the primary outcome. Given the small sample this is just a pilot study so any conclusions about other outcomes will be considered preliminary. Results will provide new evidence that may lead to consider CBT-F+MIT a treatment option for ED deserving investigations in larger trials.

ELIGIBILITY:
Inclusion Criteria:

* ED diagnosed in the past 6 months
* Seeking treatment for eating disorder
* Able to provide written, informed consent
* BMI > 18.5

Exclusion Criteria:

* Acute psychotic episode, psychotic symptoms, Bipolar I disorder; antisocial personality disorder
* Suicidal ideation
* Substance abuse
* Previous psychological intervention for other eating disorders
* Currently involved in other ongoing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q6; Fairburn & Beglin, 1994) | Change from baseline until after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A self report measure assessing eating disorders over the past 4 weeks, providing a measure of the range of severity of eating disorder features.
Eating Attitude Test (EAT-26; Garner & Garfinkel, 1979) | Change from baseline until after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A self-report measure for identifying the presence of "eating disorder risk" based on attitudes, feelings and behaviors related to eating. It assesses general eating behaviour and risky behaviours.
Clinical Impairment Assessment Questionnaire (CIA 3.0; Bohn and Fairburn, 2008). | Change from baseline until after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  a self-report measure f assessing the severity of psychosocial impairment due to eating disorder features over the past 28 days.
Binge Eating Scale (BES; Gormally et al., 1992) | Change from baseline until after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  a self-report questionnaire of the behavioral, cognitive and emotional features of objective binge eating (OBE).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI; Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983) | At baseline, after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A self-report measure of trait and state anxiety.
Beck Depression Inventory (BDI; Beck, et al., 1961) | At baseline, after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A self-report measures of depression.
Symptom Check List (SCL-90) | At baseline, after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A measure of psychopathology symptoms and their intensity at a specific point in time.
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | At baseline, after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  A self-report scale measuring individual differences in the ability to identify, accept and manage emotional experiences. This measure help in understanding emotional dysregulation that might underlie the disorders.
Structured Clinical Interview for DSM-5 Disorders (SCID-5; Michael B. First, Janet B.W. Williams) | At baseline
  For assessing and defining DSM-5 Model for Personality Disorders.
Toronto Alexithymia Scale (TAS - 20; Taylor & Bagby, 1992) | At baseline, after 10 sessions, at the end of the treatment and in the following 3, 6, 12, 18 and 24 months after the treatment.
  It assess difficulties in understanding, processing, or describing emotions
Working Alliance Inventory-Short Revised (WAI; SR Hatcher & Gillaspy, 2006) | Every 4 weeks
  It measure the therapeutic alliance by assessing three main aspects of the therapeutic alliance: agreement on the tasks of therapy, agreement on the goals of therapy and development of an affective bond.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Fioravanti, Principal Investigator — Centro di Trattamento Integrato. Disturbi Alimentari e Obesità (CTI) di Gloria Fioravanti; Raffaele Popolo, Study Director — Centro di Terapia Metacognitiva Interpersonale, Roma
Locations (1):
- Centro di Trattamento Integrato. Disturbi Alimentari e Obesità (CTI) di Gloria Fioravanti, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Yes
Outcomes, age, gender
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 10 years
Access Criteria: Someone who has a request

REFERENCES:
- [Background] Fairburn CG, Norman PA, Welch SL, O'Connor ME, Doll HA, Peveler RC. A prospective study of outcome in bulimia nervosa and the long-term effects of three psychological treatments. Arch Gen Psychiatry. 1995 Apr;52(4):304-12. doi: 10.1001/archpsyc.1995.03950160054010. PMID 7702447
- [Background] Fairburn, CG. Interpersonal psychotherapy for bulimia nervosa. 1997
- [Background] Halmi KA, Goldberg SC, Cunningham S. Perceptual distortion of body image in adolescent girls: distortion of body image in adolescence. Psychol Med. 1977 May;7(2):253-7. doi: 10.1017/s0033291700029330. PMID 877188
- [Background] Bruch, H. (1973). Psychiatric aspects of obesity. Psychiatric Annals, 3(7), 6-9.
- [Background] Bauer, B. G., & Anderson, W. P. (1989). Bulimic beliefs: Food for thought. Journal of Counseling & Development, 67(7), 416-419.
- [Background] Casper, R. C. (1983). On the emergence of bulimia nervosa as a syndrome a historical view. International Journal of Eating Disorders, 2(3), 3-16.
- [Background] Davis C. Normal and neurotic perfectionism in eating disorders: an interactive model. Int J Eat Disord. 1997 Dec;22(4):421-6. doi: 10.1002/(sici)1098-108x(199712)22:43.0.co;2-o. PMID 9356890
- [Background] Bastiani AM, Rao R, Weltzin T, Kaye WH. Perfectionism in anorexia nervosa. Int J Eat Disord. 1995 Mar;17(2):147-52. doi: 10.1002/1098-108x(199503)17:23.0.co;2-x. PMID 7757095
- [Background] Ruggiero GM, Levi D, Ciuna A, Sassaroli S. Stress situation reveals an association between perfectionism and drive for thinness. Int J Eat Disord. 2003 Sep;34(2):220-6. doi: 10.1002/eat.10191. PMID 12898558
- [Background] Vitousek, K. B., & Hollon, S. D. (1990). The investigation of schematic content and processing in eating disorders. Cognitive therapy and research, 14(2), 191-214.
- [Background] Button EJ, Loan P, Davies J, Sonuga-Barke EJ. Self-esteem, eating problems, and psychological well-being in a cohort of schoolgirls aged 15-16: a questionnaire and interview study. Int J Eat Disord. 1997 Jan;21(1):39-47. doi: 10.1002/(sici)1098-108x(199701)21:13.0.co;2-4. PMID 8986516
- [Background] Button EJ, Sonuga-Barke EJ, Davies J, Thompson M. A prospective study of self-esteem in the prediction of eating problems in adolescent schoolgirls: questionnaire findings. Br J Clin Psychol. 1996 May;35(2):193-203. doi: 10.1111/j.2044-8260.1996.tb01176.x. PMID 8773797
- [Background] Canals J, Carbajo G, Fernandez J, Marti-Henneberg C, Domenech E. Biopsychopathologic risk profile of adolescents with eating disorder symptoms. Adolescence. 1996 Summer;31(122):443-50. PMID 8726902
- [Background] Geller J, Srikameswaran S, Cockell SJ, Zaitsoff SL. Assessment of shape- and weight-based self-esteem in adolescents. Int J Eat Disord. 2000 Nov;28(3):339-45. doi: 10.1002/1098-108x(200011)28:33.0.co;2-r. PMID 10942921
- [Background] Ghaderi A, Scott B. Prevalence, incidence and prospective risk factors for eating disorders. Acta Psychiatr Scand. 2001 Aug;104(2):122-30. doi: 10.1034/j.1600-0447.2001.00298.x. PMID 11473506
- [Background] Lilenfeld LR, Kaye WH, Greeno CG, Merikangas KR, Plotnicov K, Pollice C, Rao R, Strober M, Bulik CM, Nagy L. A controlled family study of anorexia nervosa and bulimia nervosa: psychiatric disorders in first-degree relatives and effects of proband comorbidity. Arch Gen Psychiatry. 1998 Jul;55(7):603-10. doi: 10.1001/archpsyc.55.7.603. PMID 9672050
- [Background] Neumark-Sztainer D, Hannan PJ. Weight-related behaviors among adolescent girls and boys: results from a national survey. Arch Pediatr Adolesc Med. 2000 Jun;154(6):569-77. doi: 10.1001/archpedi.154.6.569. PMID 10850503
- [Background] Rastam M. Anorexia nervosa in 51 Swedish adolescents: premorbid problems and comorbidity. J Am Acad Child Adolesc Psychiatry. 1992 Sep;31(5):819-29. doi: 10.1097/00004583-199209000-00007. PMID 1400112
- [Background] Wichstrom L. Social, psychological and physical correlates of eating problems. A study of the general adolescent population in Norway. Psychol Med. 1995 May;25(3):567-79. doi: 10.1017/s0033291700033481. PMID 7480437
- [Background] Fairburn CG, Welch SL, Doll HA, Davies BA, O'Connor ME. Risk factors for bulimia nervosa. A community-based case-control study. Arch Gen Psychiatry. 1997 Jun;54(6):509-17. doi: 10.1001/archpsyc.1997.01830180015003. PMID 9193191
- [Background] Fairburn CG, Doll HA, Welch SL, Hay PJ, Davies BA, O'Connor ME. Risk factors for binge eating disorder: a community-based, case-control study. Arch Gen Psychiatry. 1998 May;55(5):425-32. doi: 10.1001/archpsyc.55.5.425. PMID 9596045
- [Background] Fairburn CG, Cooper Z, Doll HA, Welch SL. Risk factors for anorexia nervosa: three integrated case-control comparisons. Arch Gen Psychiatry. 1999 May;56(5):468-76. doi: 10.1001/archpsyc.56.5.468. PMID 10232302
- [Background] Steinberg, S., Tobin, D., & Johnson, C. (1990). The role of bulimic behaviors in affect regulation: Different functions for different patient subgroups?. International Journal of Eating Disorders, 9(1), 51-55.
- [Background] Waller, G. (2002). The psychology of binge eating. Eating disorders and obesity: A comprehensive handbook, 2, 98-102.
- [Background] Claes L, Vandereycken W, Vertommen H. Self-injurious behaviors in eating-disordered patients. Eat Behav. 2001 Autumn;2(3):263-72. doi: 10.1016/s1471-0153(01)00033-2. PMID 15001035
- [Background] Holderness CC, Brooks-Gunn J, Warren MP. Co-morbidity of eating disorders and substance abuse review of the literature. Int J Eat Disord. 1994 Jul;16(1):1-34. doi: 10.1002/1098-108x(199407)16:13.0.co;2-t. PMID 7920577
- [Background] Paul T, Schroeter K, Dahme B, Nutzinger DO. Self-injurious behavior in women with eating disorders. Am J Psychiatry. 2002 Mar;159(3):408-11. doi: 10.1176/appi.ajp.159.3.408. PMID 11870004
- [Background] Fairburn CG, Shafran R, Cooper Z. A cognitive behavioural theory of anorexia nervosa. Behav Res Ther. 1999 Jan;37(1):1-13. doi: 10.1016/s0005-7967(98)00102-8. PMID 9922553
- [Background] Steiger H, Gauvin L, Jabalpurwala S, Seguin JR, Stotland S. Hypersensitivity to social interactions in bulimic syndromes: relationship to binge eating. J Consult Clin Psychol. 1999 Oct;67(5):765-75. doi: 10.1037//0022-006x.67.5.765. PMID 10535243
- [Background] Agras WS, Walsh T, Fairburn CG, Wilson GT, Kraemer HC. A multicenter comparison of cognitive-behavioral therapy and interpersonal psychotherapy for bulimia nervosa. Arch Gen Psychiatry. 2000 May;57(5):459-66. doi: 10.1001/archpsyc.57.5.459. PMID 10807486
- [Background] Steiger H, Leung F, Thibaudeau J, Houle L, Ghadirian AM. Comorbid features in bulimics before and after therapy: are they explained by axis II diagnoses, secondary effects of bulimia, or both? Compr Psychiatry. 1993 Jan-Feb;34(1):45-53. doi: 10.1016/0010-440x(93)90035-3. PMID 8425392
- [Background] Fairburn, C. G. (2008). Cognitive behavior therapy and eating disorders. Guilford Press.
- [Background] Fairburn CG, Cooper Z, Shafran R. Cognitive behaviour therapy for eating disorders: a "transdiagnostic" theory and treatment. Behav Res Ther. 2003 May;41(5):509-28. doi: 10.1016/s0005-7967(02)00088-8. PMID 12711261
- [Background] Cooper Z, Fairburn CG. The Evolution of "Enhanced" Cognitive Behavior Therapy for Eating Disorders: Learning From Treatment Nonresponse. Cogn Behav Pract. 2011 Aug;18(3):394-402. doi: 10.1016/j.cbpra.2010.07.007. PMID 23814455
- [Background] Dalle Grave R, Calugi S, Doll HA, Fairburn CG. Enhanced cognitive behaviour therapy for adolescents with anorexia nervosa: an alternative to family therapy? Behav Res Ther. 2013 Jan;51(1):R9-R12. doi: 10.1016/j.brat.2012.09.008. Epub 2012 Oct 4. PMID 23123081
- [Background] Dalle Grave R, Calugi S, Conti M, Doll H, Fairburn CG. Inpatient cognitive behaviour therapy for anorexia nervosa: a randomized controlled trial. Psychother Psychosom. 2013;82(6):390-8. doi: 10.1159/000350058. Epub 2013 Sep 20. PMID 24060628
- [Background] Dalle Grave R, Calugi S, El Ghoch M, Conti M, Fairburn CG. Inpatient cognitive behavior therapy for adolescents with anorexia nervosa: immediate and longer-term effects. Front Psychiatry. 2014 Feb 12;5:14. doi: 10.3389/fpsyt.2014.00014. eCollection 2014. PMID 24575055
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Palmer RL, Dalle Grave R. Enhanced cognitive behaviour therapy for adults with anorexia nervosa: a UK-Italy study. Behav Res Ther. 2013 Jan;51(1):R2-8. doi: 10.1016/j.brat.2012.09.010. Epub 2012 Oct 22. PMID 23084515
- [Background] Zipfel S, Wild B, Gross G, Friederich HC, Teufel M, Schellberg D, Giel KE, de Zwaan M, Dinkel A, Herpertz S, Burgmer M, Lowe B, Tagay S, von Wietersheim J, Zeeck A, Schade-Brittinger C, Schauenburg H, Herzog W; ANTOP study group. Focal psychodynamic therapy, cognitive behaviour therapy, and optimised treatment as usual in outpatients with anorexia nervosa (ANTOP study): randomised controlled trial. Lancet. 2014 Jan 11;383(9912):127-37. doi: 10.1016/S0140-6736(13)61746-8. Epub 2013 Oct 14. PMID 24131861
- [Background] Poulsen S, Lunn S, Daniel SI, Folke S, Mathiesen BB, Katznelson H, Fairburn CG. A randomized controlled trial of psychoanalytic psychotherapy or cognitive-behavioral therapy for bulimia nervosa. Am J Psychiatry. 2014 Jan;171(1):109-16. doi: 10.1176/appi.ajp.2013.12121511. PMID 24275909
- [Background] Wonderlich SA, Peterson CB, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ. A randomized controlled comparison of integrative cognitive-affective therapy (ICAT) and enhanced cognitive-behavioral therapy (CBT-E) for bulimia nervosa. Psychol Med. 2014 Feb;44(3):543-53. doi: 10.1017/S0033291713001098. Epub 2013 May 23. PMID 23701891
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Background] Fairburn CG, Bailey-Straebler S, Basden S, Doll HA, Jones R, Murphy R, O'Connor ME, Cooper Z. A transdiagnostic comparison of enhanced cognitive behaviour therapy (CBT-E) and interpersonal psychotherapy in the treatment of eating disorders. Behav Res Ther. 2015 Jul;70:64-71. doi: 10.1016/j.brat.2015.04.010. Epub 2015 Apr 22. PMID 26000757
- [Background] Le Grange D, Eckhardt S, Dalle Grave R, Crosby RD, Peterson CB, Keery H, Lesser J, Martell C. Enhanced cognitive-behavior therapy and family-based treatment for adolescents with an eating disorder: a non-randomized effectiveness trial. Psychol Med. 2020 Dec 3;52(13):1-11. doi: 10.1017/S0033291720004407. Online ahead of print. PMID 33267919
- [Background] Frostad S, Danielsen YS, Rekkedal GA, Jevne C, Dalle Grave R, Ro O, Kessler U. Implementation of enhanced cognitive behaviour therapy (CBT-E) for adults with anorexia nervosa in an outpatient eating-disorder unit at a public hospital. J Eat Disord. 2018 May 29;6:12. doi: 10.1186/s40337-018-0198-y. eCollection 2018. PMID 29854400
- [Background] Frostad S, Calugi S, Engen CBN, Dalle Grave R. Enhanced cognitive behaviour therapy (CBT-E) for severe and extreme anorexia nervosa in an outpatient eating disorder unit at a public hospital: a quality-assessment study. J Eat Disord. 2021 Nov 2;9(1):143. doi: 10.1186/s40337-021-00499-1. PMID 34727976
- [Background] Fairburn CG, Patel V. The global dissemination of psychological treatments: a road map for research and practice. Am J Psychiatry. 2014 May;171(5):495-8. doi: 10.1176/appi.ajp.2013.13111546. No abstract available. PMID 24788281
- [Background] Linardon J, Hindle A, Brennan L. Dropout from cognitive-behavioral therapy for eating disorders: A meta-analysis of randomized, controlled trials. Int J Eat Disord. 2018 May;51(5):381-391. doi: 10.1002/eat.22850. Epub 2018 Mar 1. PMID 29493805
- [Background] Allen KL, Fursland A, Raykos B, Steele A, Watson H, Byrne SM. Motivation-focused treatment for eating disorders: a sequential trial of enhanced cognitive behaviour therapy with and without preceding motivation-focused therapy. Eur Eat Disord Rev. 2012 May;20(3):232-9. doi: 10.1002/erv.1131. Epub 2011 Jul 26. PMID 21793108
- [Background] Thompson-Brenner H, Shingleton RM, Thompson DR, Satir DA, Richards LK, Pratt EM, Barlow DH. Focused vs. Broad enhanced cognitive behavioral therapy for bulimia nervosa with comorbid borderline personality: A randomized controlled trial. Int J Eat Disord. 2016 Jan;49(1):36-49. doi: 10.1002/eat.22468. Epub 2015 Dec 9. PMID 26649812
- [Background] Semerari, A., Carcione, A., Dimaggio, G., Falcone, M., Nicolo, G., Procacci, M., & Alleva, G. (2003). How to evaluate metacognitive functioning in psychotherapy? The metacognition assessment scale and its applications. Clinical Psychology & Psychotherapy, 10(4), 238-261.
- [Background] Aloi M, Rania M, Caroleo M, Carbone EA, Fazia G, Calabro G, Segura-Garcia C. How are early maladaptive schemas and DSM-5 personality traits associated with the severity of binge eating? J Clin Psychol. 2020 Mar;76(3):539-548. doi: 10.1002/jclp.22900. Epub 2019 Nov 16. PMID 31733127
- [Background] Aloi M, Rania M, Carbone EA, Caroleo M, Calabro G, Zaffino P, Nicolo G, Carcione A, Coco GL, Cosentino C, Segura-Garcia C. Metacognition and emotion regulation as treatment targets in binge eating disorder: a network analysis study. J Eat Disord. 2021 Feb 15;9(1):22. doi: 10.1186/s40337-021-00376-x. PMID 33588943
- [Background] Monteleone, A. M., Corsi, E., Cascino, G., Ruzzi, V., Ricca, V., Ashworth, R., ... & Cardi, V. (2020). The interaction between mentalizing, empathy and symptoms in people with eating disorders: A network analysis integrating experimentally induced and self-report measures. Cognitive Therapy and Research, 44(6), 1140-1149.
- [Background] Westwood H, Kerr-Gaffney J, Stahl D, Tchanturia K. Alexithymia in eating disorders: Systematic review and meta-analyses of studies using the Toronto Alexithymia Scale. J Psychosom Res. 2017 Aug;99:66-81. doi: 10.1016/j.jpsychores.2017.06.007. Epub 2017 Jun 11. PMID 28712432
- [Background] Gilbert, P., & Leahy, R. L. (Eds.). (2009). La relazione terapeutica in terapia cognitivo comportamentale. Eclipsi.
- [Background] Boone L, Braet C, Vandereycken W, Claes L. Are maladaptive schema domains and perfectionism related to body image concerns in eating disorder patients? Eur Eat Disord Rev. 2013 Jan;21(1):45-51. doi: 10.1002/erv.2175. Epub 2012 May 3. PMID 22556040
- [Background] Meneguzzo P, Cazzola C, Castegnaro R, Buscaglia F, Bucci E, Pillan A, Garolla A, Bonello E, Todisco P. Associations Between Trauma, Early Maladaptive Schemas, Personality Traits, and Clinical Severity in Eating Disorder Patients: A Clinical Presentation and Mediation Analysis. Front Psychol. 2021 Mar 31;12:661924. doi: 10.3389/fpsyg.2021.661924. eCollection 2021. PMID 33868136
- [Background] Dimaggio, G, Semerari, A, Carcione, A, Nicolō, G, & Procacci, M. Psychotherapy of personality disorders: Metacognition, states of mind and interpersonal cycles. 2007; Routledge.
- [Background] Dimaggio G, D'Urzo M, Pasinetti M, Salvatore G, Lysaker PH, Catania D, Popolo R. Metacognitive interpersonal therapy for co-occurrent avoidant personality disorder and substance abuse. J Clin Psychol. 2015 Feb;71(2):157-66. doi: 10.1002/jclp.22151. Epub 2014 Dec 31. PMID 25557644
- [Background] Salvatore G, Buonocore L, Ottavi P, Popolo R, Dimaggio G. Metacognitive Interpersonal Therapy for Treating Persecutory Delusions in Schizophrenia. Am J Psychother. 2018 Dec 1;71(4):164-174. doi: 10.1176/appi.psychotherapy.20180039. Epub 2018 Nov 21. PMID 30458633
- [Background] Gordon-King K, Schweitzer RD, Dimaggio G. Metacognitive Interpersonal Therapy for Personality Disorders Featuring Emotional Inhibition: A Multiple Baseline Case Series. J Nerv Ment Dis. 2018 Apr;206(4):263-269. doi: 10.1097/NMD.0000000000000789. PMID 29377848
- [Background] Inchausti, F., Moreno-Campos, L., Prado-Abril, J., Sánchez-Reales, S., Fonseca-Pedrero, E., MacBeth, A., ... & Dimaggio, G. (2020). Metacognitive Interpersonal Therapy in group for personality disorders: Preliminary results from a pilot study in a public mental health setting. Journal of Contemporary Psychotherapy, 50(3), 197-203.
- [Background] Popolo R, MacBeth A, Brunello S, Canfora F, Ozdemir E, Rebecchi D, Toselli C, Venturelli G, Salvatore G, Dimaggio G. Metacognitive interpersonal therapy in group: a feasibility study. Res Psychother. 2018 Dec 18;21(3):338. doi: 10.4081/ripppo.2018.338. eCollection 2018 Dec 19. PMID 32913773
- [Background] Popolo R, MacBeth A, Canfora F, Rebecchi D, Toselli C, Salvatore G, Dimaggio G. Metacognitive Interpersonal Therapy in group (MIT-G) for young adults with personality disorders: A pilot randomized controlled trial. Psychol Psychother. 2019 Sep;92(3):342-358. doi: 10.1111/papt.12182. Epub 2018 Apr 6. PMID 29624832
- [Background] Popolo R, MacBeth A, Lazzerini L, Brunello S, Venturelli G, Rebecchi D, Morales MF, Dimaggio G. Metacognitive interpersonal therapy in group versus TAU + waiting list for young adults with personality disorders: Randomized clinical trial. Personal Disord. 2022 Nov;13(6):619-628. doi: 10.1037/per0000497. Epub 2021 Aug 12. PMID 34383540
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Fairburn, C. G., & Beglin, S. J. (2008). Eating disorder examination questionnaire. Cognitive behavior therapy and eating disorders, 309, 313.
- [Background] Garner, D. M., & Garfinkel, P. A. (1979). Eating attitudes test (EAT-26): Scoring and interpretation. EAT-26 self-test.
- [Background] Bohn, K., & Fairburn, C. G. (2008). The clinical impairment assessment questionnaire (CIA). Cognitive behavioral therapy for eating disorders, 315-317.
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Derogatis, L. R., Lipman, R. S., & Covi, L. (1977). SCL-90. Administration, scoring and procedures manual-I for the R (revised) version and other instruments of the Psychopathology Rating Scales Series. Chicago: Johns Hopkins University School of Medicine.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of psychopathology and behavioral assessment, 26(1), 41-54.
- [Background] First, M. B., Williams, J. B., Karg, R. S., & Spitzer, R. L. (2016). User's guide for the SCID-5-CV Structured Clinical Interview for DSM-5® disorders: Clinical version. American Psychiatric Publishing, Inc..
- [Background] Taylor GJ, Bagby RM, Parker JD. The Revised Toronto Alexithymia Scale: some reliability, validity, and normative data. Psychother Psychosom. 1992;57(1-2):34-41. doi: 10.1159/000288571. PMID 1584897
- [Background] Hatcher, R. L., & Gillaspy, J. A. (2006). Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy research, 16(1), 12-25.
- [Background] Semerari A, Colle L, Pellecchia G, Buccione I, Carcione A, Dimaggio G, Nicolo G, Procacci M, Pedone R. Metacognitive dysfunctions in personality disorders: correlations with disorder severity and personality styles. J Pers Disord. 2014 Dec;28(6):751-66. doi: 10.1521/pedi_2014_28_137. PMID 24689762
- [Background] Grenon R, Carlucci S, Brugnera A, Schwartze D, Hammond N, Ivanova I, Mcquaid N, Proulx G, Tasca GA. Psychotherapy for eating disorders: A meta-analysis of direct comparisons. Psychother Res. 2019 Oct;29(7):833-845. doi: 10.1080/10503307.2018.1489162. Epub 2018 Jun 29. PMID 29958509
- [Background] Dimaggio, G., Salvatore, G., MacBeth, A., Ottavi, P., Buonocore, L., & Popolo, R. (2017). Metacognitive interpersonal therapy for personality disorders: A case study series. Journal of Contemporary Psychotherapy, 47(1), 11-21.
- [Background] Inchausti F, Garcia-Poveda NV, Ballesteros-Prados A, Ortuno-Sierra J, Sanchez-Reales S, Prado-Abril J, Aldaz-Armendariz JA, Mole J, Dimaggio G, Ottavi P, Fonseca-Pedrero E. The Effects of Metacognition-Oriented Social Skills Training on Psychosocial Outcome in Schizophrenia-Spectrum Disorders: A Randomized Controlled Trial. Schizophr Bull. 2018 Oct 17;44(6):1235-1244. doi: 10.1093/schbul/sbx168. PMID 29267940
- [Background] Inchausti F, Velazquez-Basterra G, Fonseca-Pedrero E, MacBeth A, Popolo R, Dimaggio G. Metacognitive interpersonal group therapy for adolescents with avoidant personality disorder: The case of Sofia. J Clin Psychol. 2022 Aug;78(8):1579-1589. doi: 10.1002/jclp.23356. Epub 2022 Mar 31. PMID 35355266
- [Background] Cheli S, Cavalletti V, Flett GL, Hewitt PL. Perfectionism unbound: An integrated individual and group intervention for those hiding imperfections. J Clin Psychol. 2022 Aug;78(8):1624-1636. doi: 10.1002/jclp.23365. Epub 2022 Apr 29. PMID 35486835
- [Background] Anderson DA, Maloney KC. The efficacy of cognitive-behavioral therapy on the core symptoms of bulimia nervosa. Clin Psychol Rev. 2001 Oct;21(7):971-88. doi: 10.1016/s0272-7358(00)00076-3. PMID 11584518
- [Background] Murphy R, Straebler S, Cooper Z, Fairburn CG. Cognitive behavioral therapy for eating disorders. Psychiatr Clin North Am. 2010 Sep;33(3):611-27. doi: 10.1016/j.psc.2010.04.004. PMID 20599136
- [Background] Davis C, Claridge G, Fox J. Not just a pretty face: physical attractiveness and perfectionism in the risk for eating disorders. Int J Eat Disord. 2000 Jan;27(1):67-73. doi: 10.1002/(sici)1098-108x(200001)27:13.0.co;2-f. PMID 10590450
- [Background] Dimaggio, G., & Lysaker, P. H. (Eds.). (2010). Metacognition and severe adult mental disorders: From research to treatment. Routledge.
- [Background] Simonsen S, Popolo R, Juul S, Frandsen FW, Sorensen P, Dimaggio G. Treating Avoidant Personality Disorder With Combined Individual Metacognitive Interpersonal Therapy and Group Mentalization-Based Treatment: A Pilot Study. J Nerv Ment Dis. 2022 Mar 1;210(3):163-171. doi: 10.1097/NMD.0000000000001432. PMID 34710894
- [Background] Misso D, Velotti P, Pasetto A, Dimaggio G. Treating intimate partner violence with metacognitive interpersonal therapy: The case of Aaron. J Clin Psychol. 2022 Jan;78(1):50-66. doi: 10.1002/jclp.23294. Epub 2021 Dec 20. PMID 34927730
- [Background] McLaren L, Gauvin L, Steiger H. A two-factor model of disordered eating. Eat Behav. 2001 Spring;2(1):51-65. doi: 10.1016/s1471-0153(00)00023-4. PMID 15001050
- [Background] Stice, E. (1994). Review of the evidence for a sociocultural model of bulimia nervosa and an exploration of the mechanisms of action. Clinical psychology review, 14(7), 633-661.
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Fairburn CG, Peveler RC, Jones R, Hope RA, Doll HA. Predictors of 12-month outcome in bulimia nervosa and the influence of attitudes to shape and weight. J Consult Clin Psychol. 1993 Aug;61(4):696-8. doi: 10.1037//0022-006x.61.4.696. PMID 8370866
- [Background] Meyer, C., Waller, G., & Waters, A. (1998). Emotional states and bulimic psychopathology. In H. W. Hoek, J. L. Treasure, & M. A. Katzman (Eds.), Neurobiology in the treatment of eating disorders (pp. 271-287). Chichester: Wiley
- [Background] Wilson GT, Fairburn CC, Agras WS, Walsh BT, Kraemer H. Cognitive-behavioral therapy for bulimia nervosa: time course and mechanisms of change. J Consult Clin Psychol. 2002 Apr;70(2):267-74. PMID 11952185
- [Background] Maher A, Cason L, Huckstepp T, Stallman H, Kannis-Dymand L, Millear P, Mason J, Wood A, Allen A. Early maladaptive schemas in eating disorders: A systematic review. Eur Eat Disord Rev. 2022 Jan;30(1):3-22. doi: 10.1002/erv.2866. Epub 2021 Oct 12. PMID 34636456
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Basile B, Novello C, Calugi S, Dalle Grave R, Mancini F. Childhood Memories in Eating Disorders: An Explorative Study Using Diagnostic Imagery. Front Psychol. 2021 Jul 22;12:685194. doi: 10.3389/fpsyg.2021.685194. eCollection 2021. PMID 34367006

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT05503745/Prot_SAP_000.pdf